CLINICAL TRIAL: NCT06587906
Title: Postoperative Complications Following Skull Base Tumor Resection: an Observational Study
Brief Title: Postoperative Complications Following Skull Base Tumor Resection
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Other Study IDs: 2023009
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Skull Base Tumor; Postoperative Complications
MeSH Terms: conditions — Skull Base Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonary ultrasound examination — All ultrasound scans were performed by the same anaesthetists. Pulmonary ultrasound examination was performed at two time points for each patient: 20 min before starting mechanical ventilation of the lungs when patients were placed in the supine position(preoperative), 20 min after after surgery end at the time the patient was placed in the supine position (postoperative), before Intubation and after extubation Patientswere scanned in the supine position following the pulmonary ultrasound examination method The thorax was divided by the anterior axillary line, the posterior axillary line, and a horizontal line beneath nipple. Twelve intercostal spaces of each area were scanned and analysed. Aeration loss was assessedby calculating the modified LUS score that is calculated mainly using the amount of B-line The pulmonary ultrasound score of the hemithorax (0-18).

SUMMARY:
The skull base tumor is located in the deep intracranial layer and is closely related to the brain stem and intracranial nerves. The incidence of postoperative complications after skull base tumor resection is high. Therefore, the perioperative management of skull base tumor resection is challenging.

DETAILED DESCRIPTION:
1. Postoperative pulmonary complications (PPCs), always had a 11.2%-24.6% high incidence rate. Pulmonary ultrasound (LUS), as a non-invasive diagnostic tool, has high accuracy in diagnosing pulmonary complications. Compared to traditional chest X-ray examinations, pulmonary ultrasound can identify PPCs such as atelectasis and pneumothorax earlier, and it is also more accurate in diagnosing lung consolidation.With relevant literature postoperative PACU pulmonary ultrasound is used to predict the area under the PPC curve (AUC) of 0.64 in patients within 8 days after non cardiac major surgery. Through pulmonary ultrasound examination, doctors can identify high-risk patients with pulmonary complications early after surgery. In this observational study, investigators aimed to assess the occurrence of PPCs within 7 days after surgery and evaluate the accuracy of preoperative and postoperative lung ultrasound scores in predicting PPCs.
2. Patients with skull base tumors often have a high risk of postoperative lower extremity venous thrombosis due to long operation time and many postoperative complications, such as long-term bed rest. If not treated in time, lower extremity venous thrombosis can cause disability, and severe cases can cause serious consequences such as pulmonary embolism due to thrombus detachment. In this observational study, investigators aimed to prospectively collect perioperative data and the occurrence of DVT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* American Society of Anesthesiologists physical status I to III
* Undergoing elective resection of skull base tumors
* Obtaining written informed consent

Exclusion Criteria:

* Heart failure, myocarditis, pericarditis, and cardiomyopathy
* Myocardial ischemia less than 6 months old
* Severe arrhythmia
* Severe bradycardia (heart rate below 50 beats per minute)
* Unable to complete preoperative cardiac assessment
* Severe liver dysfunction (Child Pugh C-grade)
* Severe lung diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older, classified as American Society of Anesthesiologists physical status I to III, who are undergoing elective resection of skull base tumors and have obtained written informed consent will be included
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications | Postoperative 7 days
  The primary outcome was the incidence of a composite endpoint of postoperative pulmonary complicationswithin 7 days after surgery. Postoperative pulmonary complications was considered to have occurred if at least one postoperative pulmonary event was observed, such as the pneumonia, pleural effusion, respiratory failure, hypoxemia, pneumothorax, atelectasis of the lung, bronchospasm..Ultrasound scans were performed at 20 min before starting mechanical ventilation of the lungs (before intubation) and performed at 20 min after surgery (after extubation)

SECONDARY OUTCOMES:
The incidence of postoperative deep venous thrombosis | Postoperative 7 days
  Lower extremity venous ultrasound, preoperative and postoperative coagulation related values, blood routine, etc
Cardiac injury | Postoperative 7 days and 30 days
  Myocardial injury was diagnosed when available troponin concentrations exceeded generation-specific and type-specific thresholds and were apparently of ischaemic origin (ie, no other obvious cause for artifactual elevation). We used the following thresholds based on available literature at time of adjudication: 1) non-high-sensitivity (fourth-generation) troponin T ≥0.03 ng/ml2; 2) high-sensitivity troponin T ≥65 ng/L; or high-sensitivity troponin T 20-64 ng/L and an increase ≥5 ng/L from baseline3; 3) high-sensitivity troponin I (Abbott assay) is ≥75 ng/L4; 4) high-sensitivity troponin I (Siemens assay) is ≥60 ng/L5; or, 5) troponin I (other assays) greater than local 99th percentiles. Myocardial infarction diagnosis required both troponin elevation and at least one diagnostic symptom or sign.
Postoperative pain | Postoperative 2 days and 7 days
  Postoperative pain evaluated by 0-10-point numerical rating scale, with high scores indicating worse pain.
Overall complications | Postoperative 7 days and 30 days
  Surgery-related complications include cardiovascular, respiratory, pulmonary, digestive, urinary, neurological, infection, and bleeding from the surgery.
Postoperative mortality rate | Postoperative 7 days and 30 days
  Follow-up by phone or mail for patient mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China